CLINICAL TRIAL: NCT07012252
Title: Optical Coherence Tomography of the Irido-Corneal Angle Before and After Goniotomy and Trabeculotomy in Primary Congenital Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Mosaad Mohammed Zmetar, Assistant Specialist of Ophthalmology at Ministry of Health of Egypt., Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-36-2019
Record Dates: First submitted 2025-05-31; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Optical Coherence Tomography; Anterior Chamber Angle; Goniotomy; Trabeculotomy; Primary Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary congenital glaucoma group (Experimental): Infants with primary congenital glaucoma.
  Interventions: Procedure: Optical coherence tomography

INTERVENTIONS:
Procedure: Optical coherence tomography — Infants underwent optical coherence tomography.

SUMMARY:
The research aimed to improve surgical techniques and long-term outcomes by utilizing this advanced imaging technology to illuminate the structural abnormalities of the anterior segment in eyes with primary congenital glaucoma.

DETAILED DESCRIPTION:
Primary congenital glaucoma (PCG) is a rare disease, but it is responsible for 2.5%-15% of all documented cases of pediatric blindness.

The main target of the treatment of pediatric glaucoma is to control the IOP surgically. However, medical treatment could be instituted as a temporary and/or adjunctive option to maximize Intraocular pressure (IOP) control. Initial goniotomy or trabeculotomy have been detected to have high success rates. Trabeculotomy has a comparable long-term success rate in most patients of PCG. The success rate of trabeculotomy is lower in advanced or late-presenting patients.

ELIGIBILITY:
Inclusion Criteria:

* Age from 1 to 72 weeks.
* Both sexes.
* Infants with primary congenital glaucoma.

Exclusion Criteria:

* Eyes in which the angle could not be visualized by the handheld anterior segment optical coherence tomography (HH AS-OCT).
* Eyes with previous intraocular surgery.

Ages: 1 Week to 72 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Central corneal thickness | 6 months post-procedure
  Central corneal thickness was measured using handheld anterior segment optical coherence tomography (HH AS-OCT).

SECONDARY OUTCOMES:
Trabecular-iris angle | 6 months post-procedure
  Trabecular-iris angle was measured using handheld anterior segment optical coherence tomography (HH AS-OCT).
Iris thickness | 6 months post-procedure
  Iris thickness was measured using handheld anterior segment optical coherence tomography (HH AS-OCT).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.